CLINICAL TRIAL: NCT06302218
Title: Erector Spinae Plane Block vs. iPACK Block With Adductor Canal Block for Pain Management in Patients Undergoing Total Knee Replacement
Brief Title: ESPB vs iPACK+ACB in Total Knee Arthroplasty
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5/2024
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Knee Arthritis; Knee Arthropathy; Knee Osteoarthritis; Knee Pain Chronic; Knee Disease; Knee Rheumatism
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ropivacaine; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- iPACK + ACB (Active Comparator): spinal anesthesia
  + ultrasound guided iPACK (20ml 0,2% ropivacaine) with ACB (10ml 0.5% ropivacaine)
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution
- Erectro Spinae Plane Block (Active Comparator): spinal anesthesia
  + ultrasound guided ESPBk - 20ml 0,2% ropivacaine
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution
- Control group (Placebo Comparator): Only spinal anesthesia - No peripheral nerve block
  Interventions: Drug: control group

INTERVENTIONS:
Drug: Ropivacaine 0.2% Injectable Solution — iPACK block + Adductor Canal Block
  Other Names: iPACK + ACB
  Arms: iPACK + ACB
Drug: Ropivacaine 0.2% Injectable Solution — Erector Spinae Plane Block
  Other Names: ESPB
  Arms: Erectro Spinae Plane Block
Drug: control group — only spinal anesthesia
  Other Names: only spinal anesthesia
  Arms: Control group

SUMMARY:
Effect of iPACK block with Adductor Canal Block and ESPB on pain management, and NLR and PLR following knee arthroplasty

DETAILED DESCRIPTION:
Knee arthroplasty is one of the most common orthopaedic procedures, especially in elderly patients, due to the deformation of joints. Patients may complain of severe pain due to surgical trauma and prostheses. Regional anaesthesia methods may be performed to reduce the surgery's induced stress response, opioid consumption, and opioid-related side effects.

In recent years, the influence of regional anesthesiology on reducing the inflammatory response after surgical procedures has been emphasised. However, very few studies have evaluated the effect of various methods of anaesthesia on the NLR and PLR.

This is the first study to investigate the effect of regional anaesthesia on the pain managementonse expres and stress respsed by the NLR and PLR in patients undergoing knee replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA classification I-III, Aged 20-90 years, Who will be scheduled for knee arthroplasty under spinal anaesthesia.

Exclusion Criteria:

* patients who have a history of bleeding diathesis,
* take anticoagulant therapy,
* have a History of chronic pain before surgery,
* have Multiple trauma, cannot assess their pain (dementia),
* have been operated on under general anaesthesia,
* have an infection in the area and do not accept the procedure

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | 48 hours after surgery
  Total opiate consumption after surgery

SECONDARY OUTCOMES:
Time to first rescue opiate analgesia | 48 hours after procedure
  Time after surgery when the patient needs opiate for the first time
Numerical Rating Scale [range 0:10] | Time Frame: 4 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | Time Frame: 8 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | Time Frame: 12 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | Time Frame: 16 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | Time Frame: 20 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | Time Frame: 24 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | Time Frame: 36 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | Time Frame: 48 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Neutrophil-to-lymphocyte ratio | 24 hours after surgery
  Neutrophil-to-lymphocyte ratio
Neutrophil-to-lymphocyte ratio | 48 hours after surgery
  Neutrophil-to-lymphocyte ratio
Platelet-to-lymphocyte ratio | 24 hours after surgery
  Platelet-to-lymphocyte ratio
Platelet-to-lymphocyte ratio | 48 hours after surgery
  Platelet-to-lymphocyte ratio
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | Postoperative 24 hours period
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating

CONTACTS AND LOCATIONS:
Overall Officials: Łukasz Łapaj, Ph.D., Study Chair — Poznań University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poznań, Poland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 month after study completion
Access Criteria: from the corresponding author on the resonable request